CLINICAL TRIAL: NCT04806672
Title: Euthyroid Sick Syndrome (ESS)….. Can it Influence Morbidity and Mortality in Moderate to Severe Traumatic Brain Injury Patients or Correlate With Glial Fibrillary Acidic Protein (GFAP) Level.
Brief Title: Euthyroid Sick Syndrome (ESS) Effect on Traumatic Brain Injury Patients and Its Relation With GFAP Level
Acronym: ESS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Hameed Mohammed, Assistant lecturer, Minia University
Other Study IDs: 695:12/2020
Record Dates: First submitted 2021-03-14; First posted 2021-03-19 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Euthyroid Sick Syndromes in Traumatic Brain Injury Patient and GFAP Level

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Euthyroid sick syndrome (ESS) effects on patients suffering from traumatic brain injury (TBI) have received little attention. Moreover, there is limited evidence that serum levels of thyroid-related hormones might influence functional outcome in the acute phase of brain damage. However, the relationship is complex, and the relevance for functional outcome and the question of therapeutic interventions remain the subject of ongoing researches .

Historically, a wide range of brain damage markers have been examined in TBI patients. However, owing to the limited tissue specificity and other concerns, most markers, including neuro-specific enolase and S100B protein, were compromised in routine clinical use .

Glial fibrillary acidic protein (GFAP) was recently reported to have greater prognostic value than other biomarkers in TBI patients as a monomeric intermediate filament protein concentrated in the astroglial cytoskeleton; GFAP is specific to brain tissue and is not routinely found in peripheral blood circulation. However, GFAP is released after astrocyte death, making it an ideal candidate marker for brain injury patients . Several studies have found that the serum levels of GFAP on admission were significantly increased in TBI patients, also a correlation between serum concentrations and the pathological types of brain damage and clinical outcomes were also reported . However, the changes in serum GFAP over time and the associated predictive utility over the acute days post injury are largely unknown.

To study the hypothesis of euthyroid sick syndrome (ESS) traumatic brain injury patients and its relation with GFAP.

DETAILED DESCRIPTION:
After obtaining the approval of research ethical committee of faculty of medicine ,El-Minia university and taking informed written consent from the participants or their relatives, this prospective cross sectional non randomized observational study will be conducted in emergency ICU of anesthesiology and intensive care department in El-Minia university hospital ,on Patients suffering from isolated moderate to severe traumatic brain injury GCS (12-3) during the period from January2021 to December 2021. Based on inclusion and exclusion criteria, patients who met eligibility criteria, the prognosis and outcome of traumatic brain injury will be observed.

Parameters assessed:

Medical history Glasgow coma scale (GCS) on admission and daily Brain computerized tomography (CT) on admission ,3rd and 5th days Thyroid functions fT3, fT4, TSH and rT3.will be assessed on admission, after24h, 3rd and 7th days.

APACHE II score ("Acute Physiology And Chronic Health Evaluation II ") Which will be assessed in admission day

SOFA score The sequential organ failure assessment score (SOFA score), Which will be assessed every day. Glial fibrillary acidic protein (GFAP). On admission ,1st,3rd and 7th days Mechanical ventilation. Length of ICU Stay. Short term outcome after 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Age : between (18-60) years old.
* Gender : both males and females.
* Isolated moderate to severe traumatic brain injury(TBI) GCS (3-12) who is expected to survive for more than 24 hours

Exclusion Criteria:

* Poly trauma patients.
* Critically ill patients.
* Patients with history of endocrinal disturbance involving both hypothalamo-pituitary axis and thyroid gland.
* Patients receiving antithyroid medication or hormonal replacement like thyroxin and insulin.
* Pregnant and lactating females.
* Patients with history neurological or psychiatric disorders.
* Patients with liver or renal failure.
* Patients with recent use of amiodarone or β-blockers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients suffering from isolated moderate to severe traumatic brain injury GCS (12-3) during the period from January 2021 to December 2021
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence | 1year
  to investigate the incidence of euthyroid sick syndrome (ESS) in traumatic brain injury patients.
morbidity and mortality | 1year
  to investigate the influence of euthyroid sick syndrome (ESS) on morbidity and mortality in traumatic brain injury patients.

SECONDARY OUTCOMES:
Disease relations | 1year
  to examine if there is any correlation between euthyroid sick syndrome (ESS) and Glial fibrillary acidic protein (GFAP) which is a sensitive biomarker for traumatic brain injury

IPD SHARING:
Plan to Share IPD: Undecided